CLINICAL TRIAL: NCT00445263
Title: Treatment by Anti GP IIb/IIIa in the Setting of a Strategy of Early Coronarography to Patients With an Acute Coronary Syndrome Without ST Elevation
Brief Title: Comparison of Two Treatment Strategies in Patients With an Acute Coronary Syndrome Without ST Elevation
Acronym: SISCA
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Because of inclusion delay
Sponsor: Hospital Avicenne (Other)
Responsible Party: Principal Investigator, FREDERIC LAPOSTOLLE, Frédéric Lapostolle, Hospital Avicenne
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PC/AP 39-2005
Record Dates: First submitted 2007-03-07; First posted 2007-03-08 (Estimated); Results first posted 2015-02-09 (Estimated); Last update posted 2015-02-27 (Estimated); Status verified 2015-02

CONDITIONS: CORONARY DISEASE
Keywords: CORONARY DISEASE
MeSH Terms: conditions — Coronary Disease | interventions — Tirofiban; Cerebral Angiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early Invasive strategy (Experimental): Tirofiban and coronarography within 6 hours
  Interventions: Drug: TIROFIBAN; Procedure: CORONAROGRAPHY
- Delayed invasive strategy (Active Comparator): Coronarography after 6 hours
  Interventions: Procedure: CORONAROGRAPHY

INTERVENTIONS:
Drug: TIROFIBAN — intravenous infusion
  Other Names: IIb/IIIa GP inhibitor
  Arms: Early Invasive strategy
Procedure: CORONAROGRAPHY — standard procedure of coronarography
  Other Names: angiography

SUMMARY:
The acute coronary syndrome (ACS) without ST elevation is a frequent pathology. The main evolutionary risk of these patients is the coronary thrombosis and its self complications. The platelets aggregation plays a major role in the physiopathology of the ACS. The therapeutic arsenal of the anti-thrombosis essentially resting on aspirin and heparin has been reinforced lately by the inhibitors of the glycoprotein anti GP IIb/IIIa. The profit of these products in the ACS with or without ST elevation, associated or not to coronarography, has clearly been demonstrated. This profit is more marked when patients are at high risk of complications. Thus, the use of an anti GP IIb/IIIa is recommended among patients at "high risk" for whom a coronarography is planned, in the last international recommendations of the European Cardiology Society (ESC), the American Heart Association and the American College of Chest Physician. Otherwise, some authors have proposed An early invasive strategy based on coronarography with discordant results. The ideal delay of realization of this coronarography is unknown. It varies according to the studies between 2.5 hours to 48 hours. Once again, patients at high risk seem to benefit the more of such a strategy if it is set precociously.

Objective To compare an invasive strategy associating an early administration of tirofiban and a coronarography achieved in the 6 hours after the randomization to a conservative strategy in a population of high risk patients with ACS without ST elevation.

Design Multicentric, prospective, randomized study.

DETAILED DESCRIPTION:
Patient's selection Patient of more than 18 years with a ACS defined by a thoracic pain of more than 20 minutes that occurred during the last 24 hours, anomalies on EKG and one of the following criteria : diabetes; recurrence of coronary pain; precocious pain post-myocardial infarction; falling of the ST segment of > 1 mm; transient elevation of the ST segment > 1 mm; elevation of the I troponin, T troponin or CPK MB; hemodynamic instability; ventricular arrhythmia; TIMI score > 5

Therapeutic modes All patients receive : aspirin, clopidogrel, enoxaparine. Trinitrin and analgesics are at the clinician's appreciation. Besides, either they receive an anti GP IIb/IIIa: tirofiban (Agrastat®) and are oriented in cardiology to have a coronarography in the six hours or they are oriented in cardiology to receive the classical treatment, guided by the investigations searching for signs of myocardial ischemia.

ELIGIBILITY:
Inclusion Criteria:

* High risk ACS without ST elevation

Exclusion Criteria:

* Age <18 years
* Pregnancy
* Persistence of the ST elevation
* Recent left branch block
* Cardiac failure or cardiogenic shock (Kilip 3 or 4)
* Treatment by anti-vitamin K
* Contra-indication to the use of one of the following treatments: aspirin, clopidogrel, enoxaparine, anti GP IIb/IIIa (tirofiban)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2007-03; Primary Completion 2010-12 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: FREDERIC LAPOSTOLLE, MD, Principal Investigator — SAMU 93 - AVICENNE HOSPITAL; FREDERIC ADNET, PHD, Study Director — SAMU 93 - AVICENNE HOSPITAL
Locations (1):
- Samu 93 - Chu Avicenne, Bobigny, Île-de-France Region, France

RESULTS

PARTICIPANT FLOW:
Groups:
- Early Invasive Strategy: Tirofiban and coronarography within six hours
- Delayed Invasive Strategy: Coronarography after six hours
Period: Overall Study
Arm/Group | Early Invasive Strategy | Delayed Invasive Strategy
Started | 83 | 87
Completed | 83 | 86
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Early Invasive Strategy | Delayed Invasive Strategy | Total
Number analyzed (Participants) | 83 | 86 | 169
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 63.9 [55.6 to 72.5] | 66.5 [57.5 to 75.8] | 65.3 [57.1 to 75.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 23 | 48
  Male | 58 | 63 | 121
BMI [Median (Inter-Quartile Range); unit: kg/m2] | 27.0 [23.6 to 29.4] | 26.6 [24.2 to 30.4] | 26.6 [24.1 to 30.1]
Family history of CVS disease [Number; unit: participants]
  Yes | 20 | 22 | 42
  No | 63 | 64 | 127
Current smoker [Number; unit: participants]
  Yes | 44 | 41 | 85
  No | 39 | 45 | 84
Diabetes mellitus [Number; unit: participants]
  Yes | 35 | 28 | 63
  No | 48 | 58 | 106
Hypertension [Number; unit: participants]
  Yes | 50 | 51 | 101
  No | 33 | 35 | 68
Dyslipidemia [Number; unit: participants]
  Yes | 45 | 45 | 90
  No | 38 | 41 | 79
Previous MI [Number; unit: participants]
  Yes | 19 | 20 | 39
  No | 64 | 66 | 130
Previous PCI [Number; unit: participants]
  Yes | 20 | 18 | 38
  No | 63 | 68 | 131
Previous CABG [Number; unit: participants]
  Yes | 8 | 4 | 12
  No | 75 | 82 | 157
On aspirin [Number; unit: participants]
  Yes | 39 | 32 | 71
  No | 44 | 54 | 98

OUTCOME MEASURES:

1. Primary Outcome: Mortality, Myocardial Infarction and Revascularization in Emergency
Time Frame: d30
Measure: Number; unit: participants
Arm/Group | Early Invasive Strategy | Delayed Invasive Strategy
Number analyzed (Participants) | 83 | 86
participants | 2 | 21

2. Secondary Outcome: Therapeutic Failure (Well Defined) During the First 6 Hours. Clinical Evolution and Electrocardiography
Time Frame: until the exit from the hospital and at d30.
Reporting Status: Not Posted

3. Secondary Outcome: Coronarographic Criteria : TIMI Score at the Beginning and the End of the Procedure; Existence of an Intra-coronary Thrombus
Time Frame: d30
Reporting Status: Not Posted

4. Secondary Outcome: Troponin Peak. Left Ventricular Ejection Fraction Before Hospital Exit. Length of Stay in USIC and Hospital. Hemorrhagic Complications.
Time Frame: d30
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Early Invasive Strategy | Delayed Invasive Strategy
Serious Adverse Events (participants affected / at risk) | 2/83 | 1/86
Other Adverse Events (participants affected / at risk) | 0/83 | 0/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Early Invasive Strategy (N=83) | Delayed Invasive Strategy (N=86)
Major bleeding (General disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No